CLINICAL TRIAL: NCT04246814
Title: Effect of Low-level Laser Therapy in the Treatment of Diabetic Foot Ulcers: a Double-blind Randomized Controlled Trial
Brief Title: Use of Low-level Laser Therapy in the Treatment of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Piaui (Other)
Responsible Party: Principal Investigator, Vinicius Saura Cardoso, PhD Professor of the Graduate Program in Biomedical Sciences, Federal University of Piaui
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17081119.1.0000.5214
Record Dates: First submitted 2020-01-22; First posted 2020-01-29 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Diabetic Foot Ulcer; Diabetic Foot
MeSH Terms: conditions — Diabetic Foot | interventions — Bandages

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Masking will be double-blind, the volunteer and outcome assessor will not be aware of the individual allocation of participants in the intervention groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CC + dressing (Placebo Comparator): The group will receive placebo LASER application associated with Helianthus annuus oil dressing.
  Interventions: Device: CC; Procedure: Dressing
- LG1 + dressing (Active Comparator): The group will receive application of LASER Gallium Arsenide (GaAs) 904 nm 10 J/cm² associated with Helianthus annuus oil dressing.
  Interventions: Device: LG1; Procedure: Dressing
- LG2 + dressing (Active Comparator): The group will receive application of LASER Gallium Arsenide (GaAs) 904 nm 8 J/cm² associated with Helianthus annuus oil dressing.
  Interventions: Device: LG2; Procedure: Dressing
- LG3 + dressing (Active Comparator): The group will receive application of LASER Gallium Arsenide (GaAs) 904 nm 4 J/cm² associated with Helianthus annuus oil dressing.
  Interventions: Device: LG3; Procedure: Dressing

INTERVENTIONS:
Device: LG1 — Application of LASER AsGa 904nm 10 J/cm².
  Arms: LG1 + dressing
Device: LG2 — Application of LASER AsGa 904nm 8 J/cm².
  Arms: LG2 + dressing
Device: LG3 — Application of LASER AsGa 904nm 4 J/cm².
  Arms: LG3 + dressing
Device: CC — Application of placebo LASER.
  Arms: CC + dressing
Procedure: Dressing — Application of Helianthus annuus oil dressing.

SUMMARY:
Diabetes mellitus (DM) is currently an important cause of morbidity and mortality. Global estimates indicate that 382 million people live with diabetes (8.3%), and that number could reach 592 million in 2035. The diabetic foot ulcers (DFU) present as sore wounds with disintegration of the skin. The DFU affect 15% of diabetic patients. Several studies have been conducted aiming to find therapeutic strategies for the healing of DFU, among the reported therapeutic methods the Low-level Laser Therapy (LLLT) has been highlighted. The aim of this study is to investigate the effects of different doses of LLLT in the treatment of DFU. Methods: This study is characterized as a double-blind randomized clinical trial (RCT), consisting of four groups, the control group will have only dressing and placebo LLLT application and the other three groups will have dressing and real LLLT GaAs 904 nm application. Expected outcomes: to elucidate the effects of different doses of LLLT GaAs 904 nm on the treatment of DFU, beyond to identify the most effective dose.

DETAILED DESCRIPTION:
All groups will perform the same procedures twice weekly. Volunteers will be comfortable with the affected foot exposed. The diabetic foot ulcers (DFU) will be cleaned using saline solution and gauze, then the ulcer temperature will be checked using the digital infrared thermometer. Diabetic wounds will be measured and photographed at baseline and every 10 visits until the study is completed, the images will be analyzed using the ImageJ program for follow-up throughout the intervention. The DFU will be ranked according to the Wagner Scale. Afterwards the volunteers will receive LLLT application and conventional treatment in the form of Helianthus Annuus oil dressing. Both therapist and participant will be instructed on precautions to be observed when using LLLT. Goggles will be provided prior to administration. The lower cylinder of the LASER probe will be placed perpendicular to the DFU, the floor and edges of the ulcer will be irradiated using punctual and scanning techniques, respectively. Once a week blood glucose levels will be obtained for patient screening. All data will be recorded until the end of the visits in a control form prepared.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus patients with diabetic foot ulcers;
* Patients aged 18 and over.

Exclusion Criteria:

* Type 2 diabetes mellitus patients with ulcers in parts of the body other than the feet;
* Patients with infected diabetic foot ulcers.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-08-27 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2023-08-18 (Actual)

PRIMARY OUTCOMES:
Change in the ulcer area | Before intervention starts, 5th and 10th week of intervention.
  Measure of ulcer area change.
Change in complete ulcer healing | Before intervention starts, 5th and 10th week of intervention.
  Change in the percentage of complete ulcer healing.

SECONDARY OUTCOMES:
Wagner Classification | Before intervention starts, 5th and 10th week of intervention and after 1 month and after 1 month.
  Ulcer categorization according to Wagner Classification.
Blood glucose | Before intervention starts, 5th and 10th week of intervention and after 1 month and after 1 month.
  Glycemic levels.
Temperature | Before intervention starts, 5th and 10th week of intervention.
  Ulcer temperature.
Short Form-36 Health Survey questionnaire | Before intervention starts, 5th and 10th week of intervention and after 1 month and after 1 month.
  The Short Form-36 Health Survey questionnaire (SF 36) assesses quality of life and consists of 36 questions, covering 8 domains. This questionnaire has a final score from 0 to 100, in which zero corresponds to the worst general health status and 100 to the best health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Piaui, Parnaíba, Piauí, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saura Cardoso V, de Souza Lima da Silveira PR, Dos Santos CM, Miranda MB, Silva Barros AC, Veloso LC, Magalhaes AT, da Rocha RB, Hazime FA. Dose-response and efficacy of 904 nm photobiomodulation on diabetic foot ulcers healing: a randomized controlled trial. Lasers Med Sci. 2024 May 28;39(1):142. doi: 10.1007/s10103-024-04090-3. PMID 38805069
- [Derived] Cardoso VS, de Souza Lima da Silveira PR, Dos Santos CM, da Rocha RB, Hazime FA. Dose-response and efficacy of low-level laser therapy on diabetic foot ulcers healing: Protocol of a randomized controlled trial. Contemp Clin Trials. 2021 Nov;110:106561. doi: 10.1016/j.cct.2021.106561. Epub 2021 Sep 4. PMID 34487920